CLINICAL TRIAL: NCT03345329
Title: Development of a Molecular Diagnosing Platform for Relieving Periodontal Symptoms
Status: Completed | Type: Observational
Sponsor: General Biologicals Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 201506030
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Periodontal Diseases; Peri-Implantitis
MeSH Terms: conditions — Periodontal Diseases; Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontal patient
- Healthy person
- Peri-implantitis patient

SUMMARY:
More than ninety percent of adults in Taiwan are suspected to carry periodontal disease, which causes bad breath, swollen and bleeding gums, plaque and even tooth loss. Half of the patients, however, are ignorance these clinical syndromes because of no obvious pain. In this study, the investigators selected six periodontal disease-associated bacteria strains, including Porphyromonas gingivalis (Pg), Fusobacterium nucleatum (Fn), Actinobacillus actinomycetemcomitans (Aa), Tannerella forsythia (Tf), Treponema denticola (Td) and Prevotella intermedia (Pi) as diagnostic markers. Using real-time PCR and MALDI Biotyper, the investigators will establish the database of oral microorganisms in Taiwanese people, providing periodontal disease clinical markers of high-risk groups and the basis for personal medicine of therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧25
2. 3≦periodontal screening and recording≦4
3. 16 natural teeths and 6 front teeth at lesat
4. GI≧1.25
5. PI≧2

Exclusion Criteria:

1. People who have oral lesion, dental braces, denture, mouthwash allergy, or serious systemic disease
2. People who have ever eaten antibiotics and Anti-inflammatory drugs over the last 6 months
3. People who have ever eaten Immunosuppressive drugs, antiepileptic drugs, antihypertensive drugs, or anticoagulant
4. Pregnant women or the woman who eat birth control pills

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age≧25
  2. 3≦periodontal screening and recording≦4
  3. 16 natural teeths and 6 front teeth at lesat
  4. GI≧1.25
  5. PI≧2
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The change of PSR score, GI, PI, and oral bacteria strains between periodontal disease patients and healthy people after receiving periodontal therapy and using mouthwash | 9 month
  To compare the value of PSR score (0-4 point), GI (0-4 point), and PI (0-5 point) with periodontal disease patients older than 60 years of age, periodontal disease patients younger than 60 years of age and healthy people after receiving periodontal therapy and using mouthwash. Oral bacteria strains are also compared with these groups.

IPD SHARING:
Plan to Share IPD: No